CLINICAL TRIAL: NCT01513538
Title: TherapyGuide : Analysis of the Acceptance and Changes to Parameters Programming Suggested by the TherapyGuide Function
Brief Title: Analysis of the Acceptance and Changes to Parameters Programming Suggested by the TherapyGuide Function
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: TherapyGuide
Record Dates: First submitted 2012-01-11; First posted 2012-01-20 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2017-05

CONDITIONS: Bradyarrhythmia
Keywords: Pacemaker programming; Bradyarrhythmia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TherapyGuide: Patients implanted with a dual chamber pacemaker featuring the TherapyGuide function
  Interventions: Device: TherapyGuide

INTERVENTIONS:
Device: TherapyGuide — Use of TherapyGuide function to help programming the device

SUMMARY:
The technological progress allowed the development of more and more sophisticated pacemakers, widening the therapeutic indications but also meeting the physiological needs of the patient. This progress led to a more and more complex programming for the physicians. To help them set optimally the pacing parameters, physicians refer to the existing recommendations of learned societies as well as to his expertise. Manufacturers developed also algorithms integrated into pacemakers with the aim of assisting physicians in their programming.

TherapyGuide is a function which proposes a programming adapted to the psychopathological state of the patient, with a justification based on experts' consensus, clinical studies as well as on published articles.

Physicians have the choice to accept or reject the programming proposed by TherapyGuide. When rejected, there is no means to analyze the modifications brought to the proposed set of parameters. The nature, the frequency and the reasons of these modifications are not thus known.

The purpose of this study is to assess the acceptance of the TherapyGuide proposals by physicians and to identify the most frequent type of programming changes they make and their rationale.

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted with a pacemaker featuring the TherapyGuide function
* Patient more than 18 years of age.
* Patient able to sign a data release authorization form

Exclusion Criteria:

- Unwillingness or inability to provide written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with a dual chamber pacemaker featuring the TherapyGuide function
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Bouchard, Marseille, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Implanted With a Dual Chamber Pacemaker: All the enrolled patients were patients implanted with a dual chamber pacemaker with the Therapy Guide application : one-arm study.
Period: Overall Study
Arm/Group | Patients Implanted With a Dual Chamber Pacemaker
Started (Screening has been stopped after 578 patients agreed to participate to the study.) | 578
Completed | 573
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | TherapyGuide
Number analyzed (Participants) | 578
Age, Customized [Mean (Full Range); unit: years]
  Men | 77 [67 to 87]
  Women | 79 [70 to 88]
Sex/Gender, Customized [Number; unit: participants]
  Men | 347
  Women | 231
Region of Enrollment [Number; unit: participants]
  France | 578

OUTCOME MEASURES:

1. Primary Outcome: Acceptance of TherapyGuide Proposals and Typology of Programming Changes
Description: The primary objective is to assess the acceptance of the TherapyGuide proposals by the physicians.
  Acceptance will be assessed by measuring the proportion of cases where physicians programmed the set of parameters recommended by the TherapyGuide with no modifications.
Time Frame: 30 months
Measure: Number; unit: percentage of patients
Groups:
- Patients Implanted With a Dual Chamber Pacemaker: All the patients were implanted with a dual chamber pacemaker with Therapy Guide function : one-arm study.
Arm/Group | Patients Implanted With a Dual Chamber Pacemaker
Number analyzed (Participants) | 573
percentage of patients | 46

ADVERSE EVENTS:
Time Frame: No adverse event collection.
Description: No adverse event collection.
Arm/Group | Patients Implanted With a Dual Chamber Pacemaker
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No